CLINICAL TRIAL: NCT01980953
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Particle Size, Formulation, and Food on the Pharmacokinetics of GDC-0032 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Particle Size, Formulation and Food on the Pharmacokinetics of GDC-0032 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GP28619
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide

ARMS (4):
- Part 1: Food Effect (Experimental): GDC-0032 will be administered orally over 3-Treatment Period (TP) in 6-sequence as one 3 milligrams (mg) capsule in TP-A after 10 hour fasting from food, one 3 mg Phase III tablet in TP-B after 10 hour fasting from food and one 3 mg Phase III tablet in TP-C following the start of standard Food and Drug Administration (FDA) high-fat breakfast. Washout period o 14 to 20 days will be given between each TP.
  Interventions: Drug: GDC-0032 Phase III Tablet; Drug: GDC-0032 Capsule
- Part 2: Tablet Formulation Comparison (Experimental): Different formulations of tablets (Tablet A and Tablet B) of GDC-0032 will be administered orally over 2-TP having 10 hour fasting from food. Participants will receive one 3 mg Tablet A in TP-A and one 3 mg Tablet B in TP-B after 14 to 20 days washout period.
  Interventions: Drug: GDC-0032 Tablet
- Part 3: Capsule API Lot Comparison (Experimental): Two different lots of GDC-0032 active pharmaceutical ingredient (API) capsule formulation will be administered orally in crossover fashion over 2-TP to 20 participants having 10 hour fasting from food. Participants will receive one 3 mg capsule in TP-A and one 3 mg capsule in TP-B after 14 to 20 days washout period.
  Interventions: Drug: GDC-0032 Capsule
- Part 4: Tablet Relative Bioavailibity (Experimental): GDC-0032 will be administered orally in crossover fashion over 2-TP to 20 participants having 10 hour fasting from food. Participants will receive one 3 mg capsule in TP-A and one 2 mg Phase III tablet in TP-B after 14 to 20 days washout period.
  Interventions: Drug: GDC-0032 Phase III Tablet; Drug: GDC-0032 Capsule

INTERVENTIONS:
Drug: GDC-0032 Phase III Tablet — Participants will receive 2 mg or 3 mg Phase III tablet after 10 hour fasting from food.
  Arms: Part 1: Food Effect; Part 4: Tablet Relative Bioavailibity
Drug: GDC-0032 Tablet — Participants will receive 3 mg Tablet A or Tablet B formulation after 10 hour fasting from food.
  Arms: Part 2: Tablet Formulation Comparison
Drug: GDC-0032 Capsule — Participants will receive 3 mg GDC-0032 capsule formulation after 10 hour fasting from food.
  Arms: Part 1: Food Effect; Part 3: Capsule API Lot Comparison; Part 4: Tablet Relative Bioavailibity

SUMMARY:
This 4-part study will assess the effect of formulation, food, and active pharmaceutical ingredient (API) lot on the pharmacokinetics of GDC-0032 in healthy volunteers. Part 1 is an open-label, 3-period, 6-sequence study, and Parts 2, 3, and 4 are open-label 2-period crossover studies. Participants will receive single doses of GDC-0032 capsule or tablet formulation, in the fasted or fed state.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential, between 18 and 55 years of age, inclusive; females will meet the following criteria: they will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year or surgically sterile for at least 90 days.
* Body mass index (BMI) 18.5 to 32 kg/m^2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), vital signs and clinical laboratory evaluations
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at each Check-in (Day -1; does include alcohol)
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV]) and negative human immunodeficiency virus (HIV) antibody screens
* Males will either be sterile or agree to use approved methods of contraception as defined by protocol from Period 1 Check-in (Period 1, Day -1) until 90 days following the last dose of study drug

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs, except for appendectomy, hernia repair, and/or cholecystectomy
* History of alcoholism or drug addiction within 1 year prior to Period 1 Check-in (Period 1, Day -1)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* History of Type 1 or 2 diabetes mellitus and/or elevated fasting glucose (greater than [>] 120 milligrams per deciliter [mg/dL]) at baseline (as confirmed by repeat)
* History of Gilbert's Syndrome
* Evidence of malabsorption syndrome or other condition that would interfere with enteral absorption
* Inability or unwillingness to swallow pills or consume high-fat breakfast
* Use of any tobacco- or nicotine-containing products within 6 months prior to Period 1 Check-in (Period 1, Day -1) and during the entire study
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Period 1 Check-in (Period 1, Day -1) and during the entire study duration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Area Under the Concentration-Time Curve Extrapolated to Infinity (AUC0-infinity) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Maximum Plasma Concentration (Cmax) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour postdose

SECONDARY OUTCOMES:
Time to Maximum Plasma Concentration (tmax) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Apparent Terminal Elimination Rate Constant | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Apparent Terminal Elimination Constant (t1/2) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Apparent Total Clearance (CL/F) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Apparent Volume of Distribution (Vz/F) | Pre-dose (Hour 0), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 168, 192 hour post-dose
Percentage of Participants With Adverse Events | From Baseline up to approximately 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Covance Research Unit - Dallas, Dallas, Texas, United States